CLINICAL TRIAL: NCT06410638
Title: Effect of Different Exercise Capacity Tests on Intercostal Muscle Oxygenation
Brief Title: Intercostal Muscle Oxygenation During Exercise Tests
Status: Recruiting | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Assoc. Prof. Dr., Istanbul Medipol University Hospital
Other Study IDs: ICM_Moxy
Record Dates: First submitted 2024-05-04; First posted 2024-05-13 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Muscle Oxygenation
Keywords: exercise capacity test; muscle oxygenation; intercostal muscle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects
  Interventions: Diagnostic Test: Six Minute Walking Test; Diagnostic Test: Shuttle walking test

INTERVENTIONS:
Diagnostic Test: Six Minute Walking Test — It is applied in a 30 m long corridor in an indoor environment, and the distance walked by the patient in a six-minute period, oxygen saturation, heart rate, and change in dyspnea are recorded. For this, before starting the test, oxygen saturation, heart rate, arterial blood pressure and dyspnea level according to the Borg scale are recorded. The same parameters are measured again at the end of the test. The feature of this test is that the person walks at his own pace, stopping when necessary and allowing the use of oxygen. It is an exercise test that is easy to perform and well tolerated.
Diagnostic Test: Shuttle walking test — Shuttle walking test at increasing speed is an exercise test in which walk between two cones 10 m apart at an increasing speed throughout the test and each 10-meter journey between the two cones is counted as a shuttle.

SUMMARY:
The aim of our study is to determine the effects of different exercise capacity tests on intercostal muscle oxygenation and to reveal the effect of changing accessory respiratory muscle oxygenation on exercise test success.

DETAILED DESCRIPTION:
In the study, intercostal muscle oxygenation will be measured in different exercise capacity tests. A total of 32 healthy young women and men between the ages of 18-25 who meet the inclusion criteria and voluntarily agree to participate in the study will be included in the study. The cases will be randomized into 2 groups: Six minute walking test group and incremental shuttle walking test group. Heart rate, oxygen saturation, and fatigue levels will be measured with the modified Borg scale before and after the tests. During the tests, oxygen levels of the intercostal muscles will be monitored with the MOXY device. After sufficient wash out time, the groups will be crossed and different exercise tests will be applied to the cases. The result of our study will provide information about the use of intercostal muscles during different exercise tests. As a result of the study, results that can be interpreted for patient groups with circulatory system, respiratory system and physical limitations will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35
* Body Mass Index <25 kg/m²
* Participating in the study voluntarily

Exclusion Criteria:

* Being a smoker
* Presence of any systemic, orthopedic or cardiopulmonary disease that may prevent exercise tests
* Presence of any diagnosed respiratory, vascular and heart disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adults
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Muscle Oxygenation of intercostal muscles | During intervention
  The measurement will be made with the MOXY device. The device will be placed on the intercostal muscle and measurements will be taken during the exercise tests. Measured values at the beginning, end and every 1 minute will be taken and analyzed.

SECONDARY OUTCOMES:
Forced expiratory pressure in one second | Baseline
  It will be performed with Cosmed Pony Fx (Italy) desktop spirometry device.
Evaluation of blood pressure | During the intervention
  Sistolik and diastolic blood pressure will be measured with the Wrist Blood Pressure Monitor
Evaluation of heart rate | During the intervention
  It will be measured with a pulse oximeter.
Evaluation of oxygen saturation | During the intervention
  It will be measured with a pulse oximeter.
Forced vital capacity | Baseline
  It will be performed with Cosmed Pony Fx (Italy) desktop spirometry device.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided